CLINICAL TRIAL: NCT02772601
Title: The Effect of Multiple Subcutaneous Doses of Risankizumab on the Single Dose Pharmacokinetics of Cytochrome P450 Substrates (Caffeine, Warfarin, Omeprazole, Metoprolol and Midazolam) Administered Orally in an Open-label, One-sequence Trial in Patients With Plaque Psoriasis With or Without Concomitant Psoriatic Arthritis
Brief Title: This Study Tests the Effect of Risankizumab on the Metabolism in the Liver of Five Additional Drugs to Study Possible Drug Interactions in Patients With Psoriasis With or Without Psoriatic Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-007; 2015-005523-31 (EudraCT Number); 1311.36 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Psoriasis
Keywords: ABBV-066; BI 655066; risankizumab
MeSH Terms: conditions — Psoriasis | interventions — Caffeine; Warfarin; Omeprazole; Metoprolol; Midazolam; risankizumab

ARMS (1):
- All patients (Experimental)
  Interventions: Drug: Caffeine; Drug: Warfarin; Drug: Omeprazole; Drug: Metoprolol; Drug: Midazolam; Drug: Risankizumab

INTERVENTIONS:
Drug: Caffeine
Drug: Warfarin
Drug: Omeprazole
Drug: Metoprolol
Drug: Midazolam
Drug: Risankizumab
  Other Names: ABBV-066; BI 655066

SUMMARY:
To assess the influence of risankizumab on kinetics of cytochrome P450 (CYP) probe drugs as a means of predicting drug-drug interactions.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated written informed consent in accordance with GCP (Good Clinical Practice) and local legislation prior to admission to the trial and prior to any trial related procedure.
* Age 18 years to 75 years at screening
* Body mass index of 18.5 to 40.0 kg/m2 and within the weight range of 50 to 148 kg
* Male or female patients.
* If female, subject must be either postmenopausal, defined as:

  * Age > 55 years with no menses for 12 or more months without an alternative medical cause.
  * Age < 55 years with no menses for 12 or more months without an alternative medical cause AND an FSH level > 40 IU/L.

OR

* Permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Females must have negative results for pregnancy tests performed:

  * at Screening on a urine sample obtained within 30 days prior to initial study drug administration, and
  * prior to initial dosing on a serum sample obtained at the start of confinement
* Women of Childbearing Potential (WOCBP) must practice at least one of the following methods of birth control, on Study Day 1 (or earlier) through at least 140 days after the last dose of study drug.

  * Combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) associated with the inhibition of ovulation, initiated at least 1 month prior to Study Day 1.
  * Progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation, initiated at least 1 month prior to Study Day 1.
  * Bilateral tubal occlusion/ligation.
  * Vasectomized partner(s), provided the vasectomized partner has received medical assessment of the surgical success and is the sole sexual partner of the WOCBP trial participant.
  * Intrauterine device (IUD).
  * Intrauterine hormone-releasing system (IUS).
  * True abstinence: Refraining from heterosexual intercourse-when this is in line with the preferred and usual lifestyle of the subject. (Note: Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable).
* Further inclusion criteria apply.

Exclusion criteria:

* Patients with

  * non-plaque forms of psoriasis (including guttate, erythrodermic, or pustular)
  * current drug-induced psoriasis (including an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
  * active ongoing inflammatory diseases other than psoriasis that might confound trial evaluations according to investigator's judgment
* Participation in another trial with an investigational drug or device within 4 weeks or 5 half-lives (whichever is greater) prior to screening. Observational study is permitted.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the study, as assessed by the investigator
* Major surgery performed within 12 weeks prior to screening or planned within 10 months after screening (e.g. hip replacement, aneurysma removal, stomach ligation)
* Active systemic infections during the last 2 weeks (exception: common cold) prior to screening
* Chronic or relevant acute infections including HIV (Human Immunodeficiency Virus), viral hepatitis and (or) tuberculosis or evidence of tuberculosis infection as defined by a positive QuantiFERON TB (tuberculosis) test within 2 months prior to or during screening. Patients with a positive QuantiFERON TB test may participate in the study if further work up including a chest X-ray (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active tuberculosis and initiation of treatment during the conduct of this study is not needed. If presence of latent tuberculosis is established, then treatment according to local country guidelines must have been initiated and completed prior to study initiation.
* Active HBV (Hepatitis B Virus) and HCV (Hepatitis C Virus), defined as:

  * HBV: hepatitis B surface antigen (HBs Ag) positive (+),HBcAb positive or detected sensitivity on the HBV deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) qualitative test for Hepatitis B core antibody (HBc Ab);
  * HCV: HCV ribonucleic acid (RNA) detectable in any subject with anti-HCV antibody (HCV Ab).
* Positive screen for drugs of abuse, alcohol or cotinine at Screening.
* Use of known inhibitors or inducers of CYP1A2, 2C9, 2C19, 2D6 or 3A4, including dietary supplements or herbal products containing St. John's wort (Hypericum perforatum) or other known CYP inducers or inhibitors within 30 days or 5 half-lives, whichever is greater prior to study CYP cocktail probe drug administration.
* Use of grapefruits, Seville oranges (sour or bitter oranges), starfruit and their juices, quinine, tonic water, dietary/herbal supplements and inhibitors of P-glycoprotein (P-gp), breast cancer resistance protein (BCRP) and organic anion-transporting polypeptide 1B1/1B3 (OATP1B1/1B3) transporters within 14 days or 5 half-lives of the respective medication before CYP cocktail probe drug administration.
* Current smokers of nicotine containing products, including those who quit smoking less than 30 days prior to CYP cocktail probe drug administration.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of uterine cervix
* Plans for administration of live vaccines during the study period or within 6 weeks prior to screening
* Further exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
AUC0 - tz (area under the concentration-time curve) of caffeine with risankizumab in plasma over time interval from 0 to last quantifiable data point | Day 98-101
AUC0 - tz (area under the concentration-time curve) of caffeine without risankizumab in plasma over time interval from 0 to last quantifiable data point | Day 1-3
AUC0 - tz (area under the concentration-time curve) of warfarin with risankizumab in plasma over time interval from 0 to last quantifiable data point | Day 98 - 105
AUC0 - tz (area under the concentration-time curve) of warfarin without risankizumab in plasma over time interval from 0 to last quantifiable data point | Day 1-8
AUC0 - tz (area under the concentration-time curve) of omeprazole with risankizumab in plasma over time interval from 0 to last quantifiable data point | Day 98 - 100
AUC0 - tz (area under the concentration-time curve) of omeprazole without risankizumab in plasma over time interval from 0 to last quantifiable data point | Day 1-2
AUC0 - tz (area under the concentration-time curve) of metoprolol with risankizumab in plasma over time interval from 0 to last quantifiable data point | Day 98 -100
AUC0 - tz (area under the concentration-time curve) of metoprolol without risankizumab in plasma over time interval from 0 to last quantifiable data point | Day 1-3
AUC0 - tz (area under the concentration-time curve) of midazolam with risankizumab in plasma over time interval from 0 to last quantifiable data point | Day 98 - 99
AUC0 - tz (area under the concentration-time curve) of midazolam without risankizumab in plasma over time interval from 0 to last quantifiable data point | Day 1-2
Cmax (maximum measured concentration) of the analyte omeprazole without risankizumab in plasma | Day 1
Cmax (maximum measured concentration) of the analyte metoprolol with risankizumab in plasma | Day 98
Cmax (maximum measured concentration) of the analyte metoprolol without risankizumab in plasma | Day 1
Cmax (maximum measured concentration) of the analyte midazolam with risankizumab in plasma | Day 98
Cmax (maximum measured concentration) of the analyte midazolam without risankizumab in plasma | Day 1
Cmax (maximum measured concentration) of the analyte caffeine with risankizumab in plasma | Day 98
Cmax (maximum measured concentration) of the analyte caffeine without risankizumab in plasma | Day 1
Cmax (maximum measured concentration) of the analyte warfarin with risankizumab in plasma | Day 98
Cmax (maximum measured concentration) of the analyte warfarin without risankizumab in plasma | Day 1
Cmax (maximum measured concentration) of the analyte omeprazole with risankizumab in plasma | Day 98

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Mcnamee, Study Director — AbbVie
Locations (1):
- Boehringer Ingelheim Investigational Site, Berlin, Germany

REFERENCES:
- [Derived] Khatri A, Cheng L, Camez A, Ignatenko S, Pang Y, Othman AA. Lack of Effect of 12-Week Treatment with Risankizumab on the Pharmacokinetics of Cytochrome P450 Probe Substrates in Patients with Moderate to Severe Chronic Plaque Psoriasis. Clin Pharmacokinet. 2019 Jun;58(6):805-814. doi: 10.1007/s40262-018-0730-x. PMID 30574672